CLINICAL TRIAL: NCT02500628
Title: Heart Rate Variability in Response to Metformin Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Woodinville Psychiatric Associates (Other)
Responsible Party: Principal Investigator, Jon Berner MD PhD, Clinic Director, Woodinville Psychiatric Associates
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150618
Record Dates: First submitted 2015-07-11; First posted 2015-07-16 (Estimated); Results first posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Fibromyalgia; Mitochondrial Diseases; Movement Disorders; Diabetes Mellitus, Type 2
Keywords: metformin; mitochondria; complex 1; fibromyalgia; neurogenic pain; diabetes; tardive dyskinesia; heart rate variability
MeSH Terms: conditions — Fibromyalgia; Mitochondrial Diseases; Movement Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus; Tardive Dyskinesia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibromyalgia (Experimental): Fibromyalgia (subgroups: opioid responsive, opioid resistant, opioid intolerant) Metformin 500 mg orally in the morning
  Interventions: Drug: Metformin
- Antipsychotic use (Experimental): Antipsychotic use (subgroups: no side effects, dyskinesia, weight gain) Metformin 500 mg orally in the morning
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500 mg orally after baseline testing of heart rate
  Other Names: Glucophage

SUMMARY:
Diseases caused by brain energy supply defects can be innate (fibromyalgia secondary to familial mitochondrial disorders) or acquired (tardive dyskinesia or weight gain associated with prolonged antipsychotic use). Patients with these possible mitochondrial disorders will provide a baseline resting heart rate sample, ingest low-dose metformin (500 mg), and then provide an additional sample 2 hours later.

DETAILED DESCRIPTION:
Doctors need to develop tests which inexpensively and reliably evaluates brain metabolism. Current diagnostic tests sample other tissues which often run on different fuels (fats), utilize unproven and often insensitive brain imaging scanners, or sequence thousands to millions of base-pairs of DNA. All of these tests are expensive. None of these tests accurately or completely capture the interactions between the 1000s of proteins involved in brain metabolism.

The investigators suspect that mathematical analysis of the resting heart rate may provide some insight into brain metabolism. The brain controls heart rate in response to changes in blood pressure and blood gases like carbon dioxide and oxygen. Tight control of heart rate is necessary to make sure that the brain has the right mix of fuel and air. Because the brain can't respond instantly to changes in its fuel supply, this system acting as a biological carburetor has a natural oscillatory rhythm that can be monitored just like frequencies on the radio.

The investigators propose to amplify these rhythms by modestly metabolically stressing the brain with metformin, a inhibitor of complex 1 in the mitochondria.

ELIGIBILITY:
Inclusion Criteria:

EITHER chronic neurogenic pain meeting American College of Rheumatology criteria for fibromyalgia or previous/current exposure to antipsychotic medications

Exclusion Criteria:

* recent infection,
* renal failure,
* pre-existing cardiac disease,
* chronic obstructive pulmonary disease
* inability to participate in informed consent,
* lack of transport to return home from study site,
* severe fasting intolerance or hypoglycemia,
* history of stroke-alike episode,
* uncontrolled migraine or cyclic vomiting,
* diabetes on insulin or sulfonylurea,
* non-English speaker,
* medications with strong effects on baseline heart rate variability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Berner, MD PhD, Principal Investigator — Woodinville Psychiatric Associates
Locations (1):
- Woodinville Psychiatric Associates, Woodinville, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7/25/2015 to 2/21/16
Period: Overall Study
Arm/Group | Fibromyalgia | Antipsychotic Use
Started | 38 | 23
Completed | 38 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fibromyalgia: Fibromyalgia (subgroups: opioid responsive, opioid resistant, opioid intolerant) Metformin 500 mg po in AM
  Metformin: 500 mg po after baseline testing of heart rate
- Antipsychotic Use: Antipsychotic use (subgroups: no side effects, dyskinesia, weight gain) Metformin 500 mg po in AM
  Metformin: 500 mg po after baseline testing of heart rate
- Total: Total of all reporting groups
Arm/Group | Fibromyalgia | Antipsychotic Use | Total
Number analyzed (Participants) | 38 | 23 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 23 | 60
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.71 (12.15) | 47.61 (11.9) | 47.1 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 23 | 61

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability (Time Domain)
Description: ratio of the standard deviation of sampled intervals between each heart beat for ten minutes at time 1 (prior to metformin ingestion) over standard deviation of the sampled intervals between each heart beat for ten minutes at time 2 (2 hours post metformin ingestion)
Time Frame: difference pre/post metformin ingestion (2 hours)
Population: Patients with or without fibromyalgia, with or without antipsychotic use.
Measure: Mean (Standard Deviation); unit: msec/msec
Arm/Group | Fibromyalgia | Antipsychotic Use
Number analyzed (Participants) | 38 | 23
msec/msec | 0.92 (0.31) | 0.83 (0.32)
Statistical Analysis 1: Comparison: Fibromyalgia vs Antipsychotic Use; comparison between fibromyalgia and non-fibromyalgia group; Test type: Other; p = 0.77, t-test, 2 sided

2. Primary Outcome: Heart Rate Variability (Frequency Domain)
Description: total power in the frequency domain is estimated for 10 minutes prior to metformin ingestion and then divided by the total power in the frequency domain estimated for 10 minutes 2 hours after metformin ingestion. Ratio is log-transformed.
Time Frame: difference pre/post metformin ingestion (2 hours)
Population: patients with or without fibromyalgia. with or without antipsychotic use
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fibromyalgia | Antipsychotic Use
Number analyzed (Participants) | 38 | 23
ratio | -.14 (0.29) | -.24 (0.38)
Statistical Analysis 1: Comparison: Fibromyalgia vs Antipsychotic Use; Test type: Other; p = 0.27, t-test, 2 sided

3. Secondary Outcome: Number of Patients Reporting Side Effects From the Medication
Description: Patient after testing generated an unprompted list of observed side effects from the medication. Many reported none. Results were scored as the binary presence or absence of side effect
Time Frame: 2 hours after ingestion
Measure: Count of Participants; unit: Participants
Arm/Group | Fibromyalgia | Antipsychotic Use
Number analyzed (Participants) | 38 | 23
Participants | 13 | 9
Statistical Analysis 1: Comparison: Fibromyalgia; difference between fibromyalgia and non-fibromyalgia patients; Test type: Other; p = 0.92, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 hours after ingestion of metformin
Description: Patients provide an unstructured summary of possible side effects. Most reported none. Common side effects of GI distress or somnolence were scored as binary presence or absence
Arm/Group | Fibromyalgia | Antipsychotic Use
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/23
Other Adverse Events (participants affected / at risk) | 13/38 | 9/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibromyalgia (N=38) | Antipsychotic Use (N=23)
GI distress (Gastrointestinal disorders) | 5 (5) | 2 (2) — Nausea
drowsiness (Nervous system disorders) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes